CLINICAL TRIAL: NCT06722235
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Study to Evaluate Efficacy and Safety of Mezagitamab Subcutaneous Injection in Participants With Chronic Primary Immune Thrombocytopenia
Brief Title: A Study of Mezagitamab in Adults With Chronic Primary Immune Thrombocytopenia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-079-3002; 2024-514401-54-00 (EU CTIS Number); jRCT2031240667 (Registry Identifier: jRCT)
Record Dates: First submitted 2024-12-05; First posted 2024-12-09 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Immune Thrombocytopenic Purpura (ITP)
Keywords: Thrombocytopenia; TAK-079; Blood Platelet Disorders; Hematologic Diseases; Cytopenia; Purpura; Hemorrhagic Disorders; Autoimmune Diseases; Immune System Diseases; Hemorrhage; Skin Manifestations; Purpura, Thrombocytopenic, Idiopathic; Purpura, Thrombocytopenic
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Thrombocytopenia; Blood Platelet Disorders; Hematologic Diseases; Cytopenia; Purpura; Hemorrhagic Disorders; Autoimmune Diseases; Immune System Diseases; Hemorrhage; Skin Manifestations; Purpura, Thrombocytopenic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mezagitamab (Experimental): Participants will receive mezagitamab injection, SC, once weekly (QW). They will receive 8 weekly doses, followed by 8 weekly doses off, and then receive 8 more weekly doses.
  Interventions: Drug: Mezagitamab
- Placebo (Placebo Comparator): Participants will receive mezagitamab placebo-matching injection, SC, QW. They will receive 8 weekly doses, followed by 8 weekly doses off, and then receive 8 more weekly doses.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mezagitamab — Mezagitamab injection administered SC.
  Other Names: TAK-079
  Arms: Mezagitamab
Drug: Placebo — Mezagitamab placebo-matching injection administered SC.
  Arms: Placebo

SUMMARY:
Primary immune thrombocytopenia (ITP) is a condition where the immune system mistakenly destroys platelets, which are cells that help stop bleeding. This leads to a low number of platelets, making it easier to bruise or bleed. The main aim of this study is to learn whether mezagitamab, when given just under the skin (subcutaneously [SC]), is effective in keeping the platelet count of adults with ITP stable when compared to a placebo. A placebo looks like medicine but doesn't have any active ingredients in it.

The participants will be treated with mezagitamab for up to 6 months.

During the study, participants will visit their study clinic several times.

Participants who complete the TAK-079-3002 study or do not have any response to study treatment by week 16 (according to study criteria) will be given the opportunity to participate in a continuation study to receive open label mezagitamab (if they are eligible and the site is able to open the continuation study).

ELIGIBILITY:
Key Inclusion Criteria:

1. The participant has been diagnosed with ITP that has persisted for at least 12 months.
2. The participant's diagnosis of ITP is supported by a prior response to an ITP therapy (not including a thrombopoietin receptor agonist [TPO-RA]), defined as having achieved a platelet count ≥50,000/μL.
3. The participant has evidence of insufficient response or intolerance to at least 1 currently available first-line therapy for treatment of ITP (for example, corticosteroids), and at least 1 currently available second-line therapy for treatment of ITP (for example, TPO-RA, rituximab, fostamatinib, mycophenolate). Insufficient response to previous treatment is defined as failure to achieve a sustained platelet count of at least 50,000/μL or doubling of baseline platelet count after an appropriate course of prior ITP treatment. Intolerance is defined as a documented side effect causing discontinuation of the therapy.
4. The participant has a mean platelet count of <30,000/μL.
5. If the participant is receiving allowed standard-of-care treatment for ITP at screening, and continued use is intended, treatment may continue during the trial if the dose, and frequency have been stable for at least 4 weeks before receiving the first dose of IMP (i.e., Day 1), and are expected to remain stable throughout the trial.
6. If the participant is an individual with potential for pregnancy, the participant is not pregnant as confirmed by negative human chorionic gonadotropin during screening, and before the first dose of trial intervention.

Key Exclusion Criteria:

1. The participant has secondary ITP.
2. The participant has had any thrombotic or embolic event within 12 months before signing the informed consent form (ICF).
3. The participant has had a splenectomy.
4. The participant has active infection with hepatitis B virus, hepatitis C virus, or human immunodeficiency virus (HIV).
5. History of malignancy (including myelodysplastic syndrome) within 5 years of signing the ICF, except for treated non-melanoma skin cancer or cervical carcinoma in situ.
6. In the opinion of the investigator, the participant has a serious medical or psychiatric illness that could potentially interfere with the completion of treatment according to this protocol.
7. The participant has received anti-cluster of differentiation (CD)20 treatment within 12 months before screening, and either of the following applies:

   1. The last dose was received within 6 months before screening.
   2. The last dose was received between 6, and 12 months before screening, and the participant has a cluster of differentiation 19 positive (CD19+) count below the lower limit of normal.
8. The participant has received any monoclonal or polyclonal antibody for immunomodulation within 6 months before Day 1.
9. The participant has any prior exposure to mezagitamab or has been exposed to another investigational agent within 4 weeks or 5 half-lives, whichever is longer, before Day 1.
10. The participant has used anticoagulants (e.g., vitamin K antagonists, direct oral anticoagulants) within 3 weeks prior to the first dose of trial treatment.
11. The participant has received a live or live-attenuated vaccine within 4 weeks prior to the first dose of trial treatment or has any live or live-attenuated vaccine planned during the trial.
12. The participant has used the following immunosuppressive agents as specified prior to the first dose of trial treatment: alkylating agents (e.g., cyclophosphamide) within 8 weeks, vinca alkaloids (e.g., vincristine) within 4 weeks, sulfones (e.g., dapsone) within 3 weeks, antiproliferative agents: (e.g., mycophenolate mofetil, and azathioprine) within 2 weeks, and calcineurin inhibitors: (e.g., cyclosporine) within 2 weeks.
13. The participant has used intravenous immunoglobulin (IVIg), SC immunoglobulin, recombinant human thrombopoietin, anti-D immunoglobulin treatment, or efgartigimod within 4 weeks before signing the ICF or it is expected that any treatment for thrombocytopenia other than the participant's standard-of-care ITP therapy (e.g., rescue therapy, administration of blood products) may be used between screening, and Day 1.
14. The participant has a history of severe allergic or anaphylactic reactions to recombinant proteins or excipients used in the mezagitamab/placebo formulation.

Other protocol defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2027-12-28 (Estimated); Study Completion 2027-12-28 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Durable Platelet Response | Up to Week 24
  Durable platelet response is defined as platelet count greater than or equal to (≥)50,000/microliter (μL) on at least 4 of the 6 weekly platelet measurements between Weeks 19 and 24.

SECONDARY OUTCOMES:
Cumulative Number of Weeks with a Platelet Count of ≥50,000/μL | Up to Week 24
  The cumulative number of weeks in which the platelet count is ≥50,000/μL through Week 24.
Time to First Platelet Count ≥50,000/μL | Up to Week 24
The Cumulative Number of Weeks with a Platelet Count of ≥30,000/μL | Up to Week 24
  The cumulative number of weeks in which the platelet count is ≥30,000/μL, and at least doubled from baseline through Week 24.
Percentage of Participants with Complete Platelet Response | Up to Week 24
  Complete platelet response is defined as a platelet count ≥100,000/μL on at least 2 visits through Week 24.
Percentage of Participants with Platelet Response at Week 16 | Week 16
  Platelet response is defined as a platelet count ≥50,000/μL before investigational medicinal product (IMP) administration at the Week 16 visit.
Change from Baseline in the Symptoms Domain Score of the Immune Thrombocytopenia Patient Assessment Questionnaire (ITP-PAQ) at Weeks 16 and 24 | Weeks 16 and 24
  ITP-PAQ is a 44-item participant reported outcome (PRO) measure that assesses disease-specific health-related quality of life (HRQoL) that includes 10 domains: Symptoms, Fatigue/Sleep, Physical Health - Bother, Physical Health - Activity, Emotional Health - Psychological, Emotional Health - Fear, Overall Quality of Life (QoL), Social Activity, Women's Reproductive Health (including Fertility subscale, and Menstrual Symptoms subscale), and Work. The 6-item symptoms domain is scored from 0 to 100, with higher scores representing improvement of symptoms.
Percentage of Participants Receiving Rescue Therapy | Up to Week 24
Percentage of Participants with Bleeding Events | Up to Week 24
  Bleeding events are defined as Grade ≥2 in the skin domain, or Grade ≥1 in the mucosal domain, or Grade ≥1 in the organ domain, in the immune thrombocytopenia-specific bleeding assessment tool (ITP-BAT) through Week 24.
Serum Concentration of Mezagitamab During and After Intervention | Predose on Day 1 and at multiple time points post-dose up to Day 169
Number of Participants with Anti-drug Antibodies (ADA) | Predose on Day 1 and at multiple time points post-dose up to Day 169
Change in ADA Titers Over Time | Up to Day 169
Number of Participants with Neutralizing ADA | Predose on Day 1 and at multiple time points post-dose up to Day 169

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (108):
- United States (18):
  - USC Norris Comprehensive Cancer Center - Keck Medicine of USC, Los Angeles, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Georgetown University Medical Center - Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - The University of Iowa, Iowa City, Iowa
  - University Of Louisville Brown Cancer Center, Louisville, Kentucky
  - American Oncology Partners of Maryland, PA, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Massachusetts Chan Medical School, Worcester, Massachusetts
  - Duke University Hospital, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - Perelman Center for Advanced Medicine (PCAM) Hospital of The University of Pennsylvania Penn Blood Disorders Program, Philadelphia, Pennsylvania
  - Lewis Katz School of Medicine at Temple University, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - University of Washingto, Seattle, Washington
  - Versiti Wisconsin, Inc, Milwaukee, Wisconsin
- Australia (10):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Concord Repatriation General Hospital, Concord, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - University of New South Wales (UNSW) - Liverpool Hospital - Liverpool Cancer Therapy Centre, Liverpool, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Monash University - Australian Centre for Blood Diseases (ACBD), Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Perth Blood Institute, West Perth, Western Australia
- Bulgaria (5):
  - Military Medical Academy Multiprofile Hospital for Active Treatment - Sofia, Sofia, Sofia-Grad
  - Medical Center "Fama Medical", Plovdiv
  - UMHAT Sv. Ivan Rilski, Sofia
  - UMHAT SofiaMed, OOD, Sofia
  - University Multiprofile Hospital for Active Treatment - Prof. Dr. Stoyan Kirkovich AD, Stara Zagora
- China (16):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hebei
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Soochow University - Shizijie Campus, Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University - Donghu Campus, Nanchang, Jiangxi
  - Shengjing Hospital of China Medical University - Nanhu Campus, Shenyang, Liaoning
  - Shaanxi Provincial People's Hospital, Xi'an, Shaanxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Jinshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - Institute of Hematology and Blood Diseases Hospital Chinese Academy of Medical Sciences - PPDS, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Zhejiang Provincial Hospital of Chinese Medicine - Main, Hangzhou, Zhejiang
- Clinical Hospital Centar Zagreb, Zagreb, Croatia
- Queen Mary Hospital, Hong Kong, Pok Fu Lam, Hong Kong
- Italy (11):
  - Azienda Ospedaliera Universitaria Federico II, Napoli, Campania
  - Universita degli Studi di Roma La Sapienza - Umberto I Policlinico di Roma, Rome, Lazio
  - Azienda Ospedaliera Di Rilievo Nazionale E Di Alta Specializzazione Garibaldi, Catania, Sicily
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi, Bologna
  - ASST Grande Ospedale Metropolitano Niguarda - Presidio Ospedaliero Ospedale Niguarda, Milan
  - Fondazione IRCCS San Gerardo Dei Tintori, Monza
  - A.O.U. Maggiore della Carita, Novara
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata, Rome
  - AOU Citta della Salute e della Scienza di Torino, Torino
  - Azienda sanitaria universitaria Giuliano Isontina, Trieste
  - Azienda ULSS 8 Berica - Ospedale San Bortolo, Vicenza
- Japan (13):
  - Chiba Aoba Municipal Hospital, Chuo-ku, Chiba
  - Chibaken Saiseikai Narashino Hospital, Narashino-shi, Chiba
  - National Hospital Organization Mito Medical Center, Ibaraki, Higashiibaraki
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Tohoku University Hospital, Sendai, Miyagi
  - Kansai Medical University Hospital, Hirakata-shi, Osaka
  - Hematology Ohta Clinic,Shinsaibashi, Osaka, Osaka
  - Osaka University Hospital, Suita-shi, Osaka
  - Saitama Medical University Hospital, Iruma-gun, Saitama
  - The University of Tokyo Hospital, Bunkyo-ku, Tokyo
  - Nihon University Itabashi Hospital, Itabashi-ku, Tokyo
  - Tokyo Metropolitan Bokutoh Hospital, Sumida-ku, Tokyo
  - Yamanashi Prefectural Central Hospital, Kofu, Yamanashi
- Netherlands (2):
  - Erasmus Medical Center, Department of Hematology, Rotterdam, South Holland
  - Hagaziekenhuis, The Hague, South Holland
- Poland (4):
  - IN-VIVO sp. z o.o., Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Instytut Hematologii i Transfuzjologii Klinika Zaburzen Hemostazy i Chorob Wewnetrznych, Warsaw, Masovian Voivodeship
  - Pratia Onkologia Katowice - PRATIA, Katowice, Silesian Voivodeship
  - N. Copernicus Provincial MCOT in Lodz, Lodz, Łódź Voivodeship
- South Korea (7):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Kyungpook National University Hospital, Daegu
  - Seoul National University Hospital (SNUH), Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Asan Medical Center, Seoul
- Spain (5):
  - Hospital Universitario Fundacion Alcorcon, Alcorcón, Mardrid
  - Hospital General Universitario Gregorio Maranon, Madrid, Mardrid
  - Hospital Universitario 12 de Octubre, Madrid, Mardrid
  - Hospital Universitario De Salaman, Salamanca
  - Hospital Universitario Virgen del Rocio, Seville
- Turkey (Türkiye) (5):
  - Ankara University Faculty of Medicine Cebeci Hospital, Department of Hematology, Mamak, Ankara
  - Aydin Adnan Menderes University Medical Faculty-Hematology Department, Efeler, Aydın
  - Cerrahpasa Tip Fakultesi, Edirne
  - Trakya Universitesi Tip Fakultesi Hastanesi, Edirne
  - Sakarya University Education and Research Hospital, Sakarya
- United Kingdom (10):
  - University Hospitals of Leicester NHS Trust, Leicester, East Midlands
  - Southampton General Hospital, Southampton, Hampshire
  - Royal Liverpool and Broadgreen University Hospitals NHS Trust, Liverpool, Merseyside
  - Greater Glasgow Health Board, Glasgow, Scotland
  - University Hospitals of North Midlands NHS Trust, Royal Stoke University Hospital, Stoke-on-Trent, Staffordshire
  - Leeds Teaching Hospitals NHS Trust, Leeds, Yorkshire
  - Guy's Hospital - Guy's & St. Thomas NHS Foundation Trust, London
  - Barts Health NHS Trust, Royal London Hospital, London
  - University College London Hospitals, London
  - Imperial College Healthcare NHS Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/bcb48c3e8d9b4904??page=1&idFilter=TAK-079-3002